CLINICAL TRIAL: NCT05704426
Title: Arrhythmia Burden in Patients With Impulse Dynamics Optimizer Cardiac Contractility Modulation (CCM) Device Implantation: Retrospective and Prospective Evaluation
Brief Title: Arrythmia Burden in Cardiac Contractility Modulation (CCM)
Acronym: ABC
Status: Terminated | Type: Observational
Why Stopped: Study is terminated due to delays.
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro2022-0954
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Arrythmia
Keywords: Impulse Dynamics Optimizer Device; Heart failure; Cardiovascular implantable electronic device; Atrial Fibrillation; Reduced ejection fraction; Internal cardioverter defibrillator; Permanent pacemaker; Arrythmia; Cardiac Contractility Modulation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Patients with available data for 6 months before the implantation of the Optimizer implantation and at least 8 months after the implantation of the optimizer at the time the study is initiated and patients with available data for 6 months before the implantation of the Optimizer implantation, but less than 8 months of follow up after Optimizer implantation at the time of the study initiation.
  Interventions: Device: Impulse Dynamics Optimizer Device
- Prospective: Patients prior to the implantation of the Optimizer that will take place as per standard of care.
  Interventions: Device: Impulse Dynamics Optimizer Device

INTERVENTIONS:
Device: Impulse Dynamics Optimizer Device — The Impulse Dynamics Optimizer is indicated for patients with New York Heart Association (NYHA) class III congestive heart failure (CHF) with left ventricular ejection fraction (LVEF) between 25 and 45% who are not candidates for cardiac resynchronization therapy. The Optimizer device requires a minimally invasive implant by a cardiac electrophysiologist with two transvenous pacemaker wires implanted into the right ventricular septum and attached to a generator in an infraclavicular region, much like a pacemaker. The Optimizer device provides CCM through improved calcium handling and has been shown to reverse the negative remodeling of the left ventricle seen in HFrEF and improve left ventricular contractile strength.

SUMMARY:
The Impulse Dynamics Optimizer Device is a Food and Drug Administration (FDA) approved; commercially available device indicated for patients with heart failure with reduced ejection fraction (HFrEF). Many candidates of this device have a previously implanted cardiovascular implantable electronic device (CIED)- internal cardioverter defibrillator (ICD) or permanent pacemaker (PM). Patients with heart failure are at high risk for both atrial and ventricular cardiac arrhythmias.

The aim of this study is to evaluate patients for Atrial fibrillation (AF) burden episode data obtained from interrogation of their CIED 8 months or greater after Optimizer implant and compare arrhythmia burden 6 months before Optimizer Cardiac Contractility Modulation (CCM) device insertion to 8 months or greater after Optimizer insertion (after 2 month blanking period).

ELIGIBILITY:
Inclusion Criteria:

1. 1%≤AF burden≤99% in the 6 month period prior to Optimizer implant as documented the patient's CIED
2. 18 years of age or older on day of signing consent
3. Any gender
4. Functional pacemaker or ICD and using remote follow-up for their CEID
5. Not scheduled for planned catheter ablation or cardioversion
6. Ability to sign consent in English or Spanish

Exclusion Criteria:

1. Permanent atrial fibrillation
2. Pregnancy (in prospective arm only)
3. Expected survival <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective patients with the Impulse Dynamics Optimizer Device already implanted and available data for at least 6 months pre-implantation and prospective patients scheduled to have the Impulse Dynamics Optimizer Device implanted as per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Jamal, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lardizabal JA, Deedwania PC. Atrial fibrillation in heart failure. Med Clin North Am. 2012 Sep;96(5):987-1000. doi: 10.1016/j.mcna.2012.07.007. Epub 2012 Aug 17. PMID 22980060
- [Background] Verma A, Kalman JM, Callans DJ. Treatment of Patients With Atrial Fibrillation and Heart Failure With Reduced Ejection Fraction. Circulation. 2017 Apr 18;135(16):1547-1563. doi: 10.1161/CIRCULATIONAHA.116.026054. PMID 28416525
- [Background] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Background] Mosterd A, Cost B, Hoes AW, de Bruijne MC, Deckers JW, Hofman A, Grobbee DE. The prognosis of heart failure in the general population: The Rotterdam Study. Eur Heart J. 2001 Aug;22(15):1318-27. doi: 10.1053/euhj.2000.2533. PMID 11465964
- [Background] Saltzman HE. Arrhythmias and heart failure. Cardiol Clin. 2014 Feb;32(1):125-33, ix. doi: 10.1016/j.ccl.2013.09.005. Epub 2013 Oct 18. PMID 24286583
- [Background] Kuschyk J, Falk P, Demming T, Marx O, Morley D, Rao I, Burkhoff D. Long-term clinical experience with cardiac contractility modulation therapy delivered by the Optimizer Smart system. Eur J Heart Fail. 2021 Jul;23(7):1160-1169. doi: 10.1002/ejhf.2202. Epub 2021 May 17. PMID 34002440
- [Background] Piccini JP, Dufton C, Carroll IA, Healey JS, Abraham WT, Khaykin Y, Aleong R, Krueger SK, Sauer WH, Wilton SB, Rienstra M, van Veldhuisen DJ, Anand IS, White M, Camm AJ, Ziegler PD, Marshall D, Bristow MR, Connolly SJ; Genotype-Directed Comparative Effectiveness Trial of Bucindolol and Toprol-XL for Prevention of Atrial Fibrillation/Atrial Flutter in Patients with Heart Failure Trial Investigators*. Bucindolol Decreases Atrial Fibrillation Burden in Patients With Heart Failure and the ADRB1 Arg389Arg Genotype. Circ Arrhythm Electrophysiol. 2021 Aug;14(8):e009591. doi: 10.1161/CIRCEP.120.009591. Epub 2021 Jul 16. PMID 34270905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retrospective
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Retrospective
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 80 [75 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Atrial Fibrillation (AF) Burden
Description: Compare the AF burden noted 6 months pre Optimizer implant to 6 post Optimizer months (post Optimizer months 3-8), after 2 month blanking period
Time Frame: 8 months post optimizer implantation
Population: AF burden was defined as the average minutes of AF/day. Outcome is reported at the pre implantation (pre-ccm) and at 6 months post (post ccm),
Measure: Mean (Full Range); unit: average minutes of AF/day
Arm/Group | Retrospective
Number analyzed (Participants) | 2
average minutes of AF/day
  pre ccm | 19.5 [15.3 to 23.6]
  post ccm | 10.2 [8.7 to 11.6]

ADVERSE EVENTS:
Description: N/A There are no adverse events as participants were not assigned to an intervention for study purposes. Only data collected for the retrospective cohort was reviewed.
Arm/Group | Retrospective
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated after only two patients in the retrospective cohort were included. No study activities were conducted for the prospective cohort and there was no formal statistical analysis conducted given the very limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT05704426/Prot_SAP_000.pdf